CLINICAL TRIAL: NCT04904926
Title: Investigating Loss of Neuromuscular Junction Transmission Fidelity in Older Adults
Acronym: STAMINA
Status: Completed | Type: Observational
Sponsor: NMD Pharma A/S (Industry)
Collaborators: Ohio University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: Sarcopenia Observational
Record Dates: First submitted 2021-05-10; First posted 2021-05-27 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Sarcopenia
Keywords: Neuromuscular Junction Transmission; Neuromuscular Disease; Repetitive Nerve Stimulation; Single Fiber EMG
MeSH Terms: conditions — Sarcopenia; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older Individuals
- Healthy young to middle aged Individuals

SUMMARY:
Sarcopenia is a condition characterised by age-related loss of muscle mass and function. Factors affecting the strength of muscle contraction independent of mass, such as neuromuscular junction (NMJ) transmission, are increasingly suspected as important contributors to the development of age-related physical disability. The group of investigators leading the current study, have recently demonstrated NMJ transmission deficits in aged mice, but whether this translates in older human individuals is not known

The primary aim is to assess whether clinically meaningfull muscle weakness is associated with NMJ transmission deficits in older human individuals with clinically meaningfull muscle weakness.

The secondary aim is to assess whether NMJ transmission deficits correlate with different measures of functional capacity to inform future trials of the most appropriate choice of tests.

DETAILED DESCRIPTION:
The study is a cross-sectional pilot study and will be led by investigators:

1. Professor Brian Clark, PhD, Ohio University
2. Professor William David Arnold, MD, Ohio State University

Up to 16 older (>70 yrs.) individuals and 8 healthy younger (18-50 yrs.) individuals will be included in this cross-sectional pilot study. To assess whether clinically meaningfull muscle weakness is associated with NMJ transmission failure, results from single fiber EMG analyses and repetitive nerve stimulation in older individuals with clinically meaningfull muscle weakness will be compared to those obtained in older adults without muscle weakness and with healthy young individuals. To assess whether NMJ transmission deficits correlates with different measures of functional capacity, a series of different functional tests will be performed.

ELIGIBILITY:
Inclusion Criteria

* Men and women 70+ years of age OR men and women 18-50 years old
* Body mass index between 19 and 40 kg/m2.
* Willingness to undergo all testing procedures, maintain current diet during the study period, and adhere to the study protocol.

Exclusion Criteria:

* Neuromuscular Disease (ie. movement disorder, or overt neurological disease, such as Sensory Neuropathy with Sensory Ataxia, Apraxia, Post-Polio Syndrome, Mitochondrial Myopathy, Myelopathy, myasthenia gravis)
* Neurological Disease (ie. Dementia (Alzheimers, multi-infarct, fronto-temporal); multiple sclerosis, amyotrophic lateral sclerosis, Parkinsons Disease, cerebellar ataxia, or significant cognitive impairment (a score of 22 or less on the Montreal Cognitive Assessment (MOCA))
* Musculoskeletal disorders (ie. rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, acute gout or osteoarthritis limiting mobility)
* Terminal illness(i.e., Cancer, myeloma, acute leukaemia)
* Uncontrolled Psychiatric disorder (ie. bipolar, schizophrenia, major depression)
* Cardiovascular Diseases (ie. NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, uncontrolled atrial fibrillation, use of a cardiac defibrillator, or uncontrolled angina or hypertension)
* Other significant conditions (ie, that would impact safety and/or compliance to the protocol (e.g. chronic renal failure requiring peritoneal or hemodialysis, chronic liver disease, blood dyscrasia, carcinoma within last 3 years, severe inflammatory bowel disease, severe respiratory disease (uncontrolled asthma, COPD), etc)
* Drug or alcohol abuse
* Not meeting MRI eligibility (e.g. metal implants, reported pregnancy or positive pregnancy test at the time of imaging for women aged 55 years or younger);
* Not meeting the DEXA eligibility (e.g. reported pregnancy or positive pregnancy test at the time of imaging for women aged 55 years or younger);
* Failure to provide informed consent;
* Subjects who do not answer "male" or female" to the question of biological sex
* Currently or recently (within the last 1 year) taking gender affirming hormones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study candidates will be referred by community physicians and other local health care providers or self-referred. Local advertising will be used to raise awareness of the study. Specifically, subjects will be recruited in one of the following ways:
  1. Through short presentations about the research project made in classes or at local community events.
  2. Email to the university community and/or the OMNI database soliciting potential volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Single Fiber Electromyography (sfEMG) | Baseline
  sfEMG of the vastus lateralis will be performed to ascertain NMJ transmission at a minimum of 30 synapses per participant.

SECONDARY OUTCOMES:
Repetitive Nerve Stimulation | Baseline
  As additional measures of NMJ transmission, Repetitive Nerve Stimulation (3Hz) of the spinal accessory nerve (recorded from the trapezius) and fibular nerve (recorded from tibialis anterior) will be performed
Magnetic Resonance Imaging | Baseline
  Assessment of thigh muscle cross-sectional area
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  Assessment of appendicular lean mass
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  Assessment of total lean mass
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  Assessment of total mass
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  ND Upper Thigh Lean Mass
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  Assessment of bone mineral density
Dual Energy X-ray Absorption (DEXA) Scanning | Baseline
  Assessment of percent body fat
Short Physical Performance Battery (SPPB) | Baseline
  Total Short Physical Performance Battery test score ranging from 0 (worst performance) to 12 (best performance)
Short Physical Performance Battery (SPPB) - Chair Stand Test | Baseline
  Chair Stand Test score ranging from 0 (worst performance) to 4 (best performance)
Short Physical Performance Battery (SPPB) - Standing Balance Test | Baseline
  Standing Balance Test score ranging from 0 (worst performance) to 4 (best performance)
Short Physical Performance Battery (SPPB) - 4 Meter Walk Test | Baseline
  4 Meter Walk Test score ranging from 0 (worst performance) to 4 (best performance)
Stair Climb Power Test | Baseline
  Assessment of lower leg power
Hand Grip Dynamometry | Baseline
  Assessment of Hand Grip Strength
Four Square Test | Baseline
  Assessment of coordination
Isometric and Isokinetic Leg Extension Strength | Baseline
  Assessment of isometric and isokinetic leg extonsor strength. Isokinetic leg extensor strength is also used for weakness classification in older adults
60-Sec MVC Fatigue Test | Baseline
  Assessment of lower extremity fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Brian Clark, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No